CLINICAL TRIAL: NCT07215169
Title: The Effect of Manual Lymph Drainage for Cancer Treatment-related External Lymphedema in the Head and Neck - a Pilot and Feasibility Study of a Randomized Controlled Trial
Brief Title: Manual Lymph Drainage for External Lymphedema
Acronym: MLD-HN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Lund University Hospital (Other)
Responsible Party: Principal Investigator, Eva Ekvall-Hansson, Professor, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023-04456-01
Record Dates: First submitted 2025-10-02; First posted 2025-10-10 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Lymphedema of Face; Neoplasms; Radiotherapy Side Effect; Lymphedema Due to Radiation
Keywords: Head and neck lymphedema management
MeSH Terms: conditions — Neoplasms; Radiation Injuries

STUDY DESIGN:
Intervention Model Description: Pilot and feasibility study of a randomized controlled trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The person who will do the randomization, the outcome assessor, and the care provider will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIT (Experimental): High-intensity treatment with manual lymphedema drainage.
  Interventions: Other: HIT
- LIT (Other): Low-intensity treatment with manual lymphedema drainage, which is the standard treatment.
  Interventions: Other: LIT

INTERVENTIONS:
Other: HIT — Manual Lymph Drainage 20 completions, first over the neck, then the face, and finally the neck again. This is repeated every second hour during the daytime.
  Arms: HIT
Other: LIT — Manual Lymph Drainage 20 completions, first over the neck, then the face, and finally the neck again once a day.
  Arms: LIT

SUMMARY:
This study will evaluate the feasibility of a randomized controlled trial. The future randomized controlled trial will compare two groups following different intensities of manual lymphatic drainage for external head- and neck lymphedema among persons treated with radiotherapy for head- and neck cancer.

DETAILED DESCRIPTION:
Methods Study setting The study will be conducted at the Department of Otorhinolaryngology, Head & Neck Surgery, Skåne University Hospital, Lund, Sweden, a tertiary referral hospital. All head and neck cancer patients in the Southern Health Care region, with a catchment area of approximately 1.2 million inhabitants, are treated at Skåne University Hospital. The patients will be assessed by the study coordinator to be able to follow and complete the intervention.

Recruitmenthttps://register.clinicaltrials.gov/prs/beta/studies/S000EE8A00000009/protocol/conditions?edit=true As part of clinical routine, the patients have a doctor´s visit three months after cancer treatment completion at the Dept. of ORL-HNS Skåne University Hospital, Lund. The assessment of lymphedema will be performed as a part of the clinical examination. Patient who are assessed to have lymphedema (>2 SD of healthy reference values13) and are possible candidates for enrolment will receive oral and written information about the study. If the patient accepts inclusion, a signed consent will be retrieved.

Intervention A: HIT

Highly Intensive Treatment with Self MLD:

Week 1 - 2: 20 strokes at the neck, 20 strokes at the cheek and finally 20 strokes at the neck, at both sides of the neck and face. This treatment should by repeated every two hours during the daytime, approximately 6-8 times a day.

Week 3 - 12: 20 strokes at the neck, 20 strokes at the cheek and finally 20 strokes at the neck, at both sides of the neck and face, once a day.

Intervention B: LIT

Low Intensive Treatment with Self MLD:

Week 1 - 12: 20 strokes at the neck, 20 strokes at the cheek and finally 20 strokes at the neck at both sides of the neck and face, once a day.

Procedure Each participant will receive a study number in order of inclusion. The code key, connecting the personal identity number with the study number, will be kept on aUSB memory stick and securely locked in at the Dept. of ORL-HNS Skåne University Hospital, Lund. Only the researchers mentioned above will have access to the code key.

Data will be retrieved from the medical records and transferred to a digital case report form (CRF)/file. BMI, measurement of tissue water data, and LyQLI questionnaires will be available as physical CRF. Each CRF will be connected to the patient's informed consent and kept securely locked as above. The data on the physical CRF will be transferred to the digital file as above. Data management will be performed according to GDPR 14.

Measurement of tissue water is performed with a lymph scanner (MoistureMeterD) at four measuring point in the head and neck area (table 1). In addition, the neck circumference at three levels will be assessed with a measuring tape (table 2). The assessments will be performed 2 and 12 weeks after interventional therapy. The measurement will be completed by a physiotherapist with specific education of HNL and the handling of the lymph scanner.

Each participant will respond to a lymphedema specific quality-of-life questionnaire, LyQLi, at the same time points as the measurements of tissue water and circumference measurements. The participants will also complete a treatment diary.

Outcomes Feasability outcomes Feasibility of a randomized controlled trial, studying the effect of Self MLD of different intensity over time for persons treated with (chemo)radiotherapy with curative intent for an oropharyngeal cancer.

The change of tissue water and neck circumference in the head and neck area at 2 weeks and 12 weeks after interventional therapy.

Patient related outcomes The difference in QoL, with specific regards to lymphedema, before and after interventional therapy.

Data collection methods

Baseline data are extracted from medical records and include:

* Diagnosis: subsite and histology type, TNM-classification, stage
* Age at diagnosis
* Gender
* BMI
* Smoking habits
* Ratings of physical activity according to Frändin and Grimby

At 14 days and 10 weeks after interventional therapy:

* BMI/weight
* Smoking habits
* Tissue water measurement in the head and neck in a sitting position
* Ratings of physical activity according to Frändin and Grimby
* Treatment diary Data analysis 40 patients (20 in each group) will be included in the study. We expect approximately 2/3 of the patients to be male according to the epidemiology of HNC.

Demographic data will be presented with medians and IQR and/or means and standard deviations (continuous variables) or numbers and percent (categorical variables).

ANOVA will be used to evaluate differences between the groups regarding the change in HNL. Wilcoxon signed rank test will be used to evaluate the differences in health related QoL with specific regards to lymphedema before and after the intervention.

Ethics and dissemination Participation in the study is voluntary. All participants can, whenever they want and without leaving any explanation, withdraw their participation. The study does not contain any physical intervention and there is no risk for harm, neither physical nor mental. The study will be performed in accordance with the ethical standards of the responsible committee on human experimentation, the Declaration of Helsinki 15.

Informed consent will be collected by Agneta Hagren and securely stored, see above.

Only the researchers mentioned above will have access to the final trial data set. The results from the study will be published in a peer-reviewed medical journal. Furthermore, the results will be communicated to the participating patients and the head and neck cancer patients' association in Sweden.

ELIGIBILITY:
Inclusion Criteria:

* • a previous diagnosis of oropharyngeal cancer (all histological types are accepted)

  * curative treatment with (chemo)radiotherapy to at least 68Gy at the primary site completed no more than 1 year before the study inclusion
  * age >18 years
  * ability to give written and informed consent.

Exclusion Criteria:

* • pregnancy

  * surgery or Botox injections in the tissue of the head and neck area
  * Locoregional deep infection i.e., suspected abscess at the scheduled time points for measurements.
  * prior daily treatment with Self MLD
  * other treatment of head and neck lymphedema, for example compression
  * psychiatric disorders
  * substance abuse problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate, retention rate, adverse events, and ability to collect outcomes | Two and twelve weeks after inclusion
  of recruitment rate, calculated as the percentage of individuals who agreed to be in the study among those who were qualified; retention rate, calculated as the percentage of individuals who completed the intervention; the ability to collect data, calculated as the percentage of completed collected data at baseline and follow-up; and adverse events, which is the num-ber of harmful or negative events that may have influenced the study procedure

CONTACTS AND LOCATIONS:
Overall Officials: Eva Ekvall Hansson, Professor, Principal Investigator — Lund University, Medical Faculty, Dep of Health Sciences
Locations (1):
- Lund university, Lund, Skåne County, Sweden